CLINICAL TRIAL: NCT05192915
Title: Comparison of Conventionally Manufactured Lower Leg Orthoses and Modular Customized Lower Leg Orthoses (AFO 4.0) in Patients With Limited Neuromuscular Foot Function During Overground Walking
Brief Title: Comparison of Conventionally Manufactured AFO and Modular Customized AFO
Acronym: AFO4-0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beat Göpfert (Other)
Responsible Party: Sponsor-Investigator, Beat Göpfert, MEng, EMBA, University of Basel
Organization: University of Basel (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AFO4-0
Record Dates: First submitted 2021-12-13; First posted 2022-01-14 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2022-11

CONDITIONS: Gait, Drop Foot
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: This study is a prospective, cross-sectional within-subjects comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modular customized AFO (Other): Walks better at self selected speed with a modular customized AFO than with a conventional AFO.
  Interventions: Device: Modular customized AFO

INTERVENTIONS:
Device: Modular customized AFO — Walks better at self selected speed with a modular customized AFO than with a conventional AFO.

SUMMARY:
The Investigator will investigate the difference in the gait pattern between 2 commercially available ankle foot orthoses (AFO): a) conventionally manufactured AFO and b) modular customized AFO using Industry 4.0 technology.

Measurement method: The participants perform an instrumented gait analyses while overground walking at a self - selected speed using a conventionally manufactured AFO or a modular customized AFO.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common movement disorder in children [Stavsky, 2017]. It is frequently accompanied by spasticity [Baker, 2009]. The typical symptoms of spastic cerebral palsy are gait abnormalities such as equinus and drop foot that lead to severe impairments in daily life [Armand, 2016]. As these symptoms will persist in adulthood, an AFO is frequently required in this patient population.

Furthermore, other neurological diseases e.g stroke [Choo, 2021], spinal cord injury, and peripheral nerve injury may require the daily use of an AFO.

Ankle-foot orthoses (AFO) have been suggested to improve the dynamic efficiency of the gait. In addition, a positive effects on gait kinetics and kinematics have been reported [Figueiredo, 2008].

Recently, modular customized AFO are increasingly proposed as their response can be tuned to the patient's gait characteristics and/or functional maturity [6]. However, the evidence on this topic is still lacking and modular customized AFO are not yet established in clinical routine.

The aim of this study is to assess gait parameters with an instrumented gait analysis of the modular customized AFO compared to conventional, untuned AFO in a group of adolescents and a group of adults using for there daily activity an AFO, while over ground walking at self selected speed over a distance of about 10 m.

ELIGIBILITY:
Inclusion Criteria:

Participants fulfilling all of the following inclusion criteria are eligible for the study:

* Patients (11-18 yrs.), who need a new orthosis (visit to an orthopedic technician)
* Patients (18-65 yrs.), who need a new orthosis (visit to an orthopedic technician)
* Informed Consent provided as documented by signature
* Confirmed diagnosis of cerebral palsy
* Confirmed diagnosis of spastic equinus and/ or drop foot,
* Gait pathologies treated with conventional AFO
* Gross Motor Function Classification System (GMFCS) level I or II

Exclusion Criteria:

* Other neuromuscular diseases
* Surgical intervention lower extremities past 12 months to improve gait pathologies
* Injections of Botulinum toxin 6 months prior to study inclusion
* Inability or unwillingness to follow the procedures of the gait analysis
* in women: pregnancy

Ages: 11 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Gait Profile Score (GPS) | immediately after the intervention (gait analysis)
  The primary outcome measure is the gait profile score (GPS), which is an overall score calculated from all kinematic parameters (joint rotation angles) of the affected leg and expressed as the deviation from the normal gait cycle in degrees.
  The outcome of the GPS will be compared between the conventional AFO, and modular customized AFO for each participant and for each group.

SECONDARY OUTCOMES:
Movement Analysis Profile (MAP) and spatial-temporal parameters | immediately after the intervention (gait analysis)
  Secondary outcomes are the Movement analysis profile (MAP) and spatial-temporal parameters, both calculated from kinematic parameters and expressed as the deviation from the normal gait cycle in degrees.
  The MAP consists of individual scores for each joint rotation angle (pelvic tilt, pelvic obliquity, pelvic rotation, hip flexion/extension, hip abduction/adduction, hip rotation, knee flexion/extension, ankle dorsiﬂexion/extension and foot progression) of the affected leg [2]. Spatial-temporal parameters are walking speed (m/s), cadence (steps/min x 100) and stride length (m) of the affected leg.
  The above-mentioned parameters will be compared between the conventional AFO, and modular customized AFO for each participant and for each group.

CONTACTS AND LOCATIONS:
Overall Officials: Beat Goepfert, MEng, EMBA, Principal Investigator — University of Basel
Locations (1):
- University of Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stavsky M, Mor O, Mastrolia SA, Greenbaum S, Than NG, Erez O. Cerebral Palsy-Trends in Epidemiology and Recent Development in Prenatal Mechanisms of Disease, Treatment, and Prevention. Front Pediatr. 2017 Feb 13;5:21. doi: 10.3389/fped.2017.00021. eCollection 2017. PMID 28243583
- [Background] Baker R, McGinley JL, Schwartz MH, Beynon S, Rozumalski A, Graham HK, Tirosh O. The gait profile score and movement analysis profile. Gait Posture. 2009 Oct;30(3):265-9. doi: 10.1016/j.gaitpost.2009.05.020. Epub 2009 Jul 24. PMID 19632117
- [Background] Armand S, Decoulon G, Bonnefoy-Mazure A. Gait analysis in children with cerebral palsy. EFORT Open Rev. 2016 Dec 22;1(12):448-460. doi: 10.1302/2058-5241.1.000052. eCollection 2016 Dec. PMID 28698802
- [Background] Choo YJ, Chang MC. Effectiveness of an ankle-foot orthosis on walking in patients with stroke: a systematic review and meta-analysis. Sci Rep. 2021 Aug 5;11(1):15879. doi: 10.1038/s41598-021-95449-x. PMID 34354172
- [Background] Figueiredo EM, Ferreira GB, Maia Moreira RC, Kirkwood RN, Fetters L. Efficacy of ankle-foot orthoses on gait of children with cerebral palsy: systematic review of literature. Pediatr Phys Ther. 2008 Fall;20(3):207-23. doi: 10.1097/PEP.0b013e318181fb34. PMID 18703958